CLINICAL TRIAL: NCT01113294
Title: Catheter Ablation for Atrial Fibrillation: A Multicenter Clinical Trial
Brief Title: Efficacy and Safety Study of Catheter Ablation for Atrial Fibrillation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuhan University (Other)
Collaborators: Peking Union Medical College (Other); Shanghai Chest Hospital (Other); Nanjing Medical University (Other); West China Hospital (Other); Guangdong Provincial People's Hospital (Other); Dalian Medical University (Other); Capital Medical University (Other)
Responsible Party: Cong-xin Huang, Renmin hospital of Wuhan university
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFCT001
Record Dates: First submitted 2010-04-21; First posted 2010-04-29 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2009-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ablation (Experimental)
  Interventions: Procedure: catheter ablation

INTERVENTIONS:
Procedure: catheter ablation — circumferential pulmonary vein isolation complex fractionated atrial electrograms ablation circumferential pulmonary vein isolation combined left atrial roof ablation circumferential pulmonary vein isolation combined left atrial isthmus ablation circumferential pulmonary vein isolation combined left atrial roof and isthmus ablation circumferential pulmonary vein isolation combined complex fractionated atrial electrograms ablation

SUMMARY:
To compare the efficacy of different procedures, identify the optimal procedure, ablation sites, ablation endpoints and post-operative anticoagulation strategy, establish the optimal treatment strategy for atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation recorded by ECG or Holter;
2. Age: 18 ~ 75 years;
3. Patients who are willing to enroll in the trial

Exclusion Criteria:

1. Patients accompanied hyperthyroidism;
2. Patients with sever liver or renal dysfunction;
3. Patients with sever cardiac dysfunction;
4. Patients had previous radiofrequency catheter ablation in the LA or Maze surgical procedure;
5. Patients with emboli in atrium;
6. Pregnant woman

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2040 (Estimated)
Dates: Start 2009-01; Primary Completion 2012-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
recurrence of atrial arrhythmias (AF, AFL, AT) | 1 month
recurrence of atrial arrhythmias (AF, AFL, AT) | 3 month
recurrence of atrial arrhythmias (AF, AFL, AT) | 6 month
recurrence of atrial arrhythmias (AF, AFL, AT) | 12 month

SECONDARY OUTCOMES:
Number of participants with all-cause death | 1 month
Number of participants with all-cause death | 3 month
Number of participants with all-cause death | 6 month
Number of participants with all-cause death | 12 month
severe blooding complications | 1 month
severe blooding complications | 3 month
severe blooding complications | 6 month
severe blooding complications | 12 month
cardio-cerebrovascular complications | 1 month
cardio-cerebrovascular complications | 3 month
cardio-cerebrovascular complications | 6 month
cardio-cerebrovascular complications | 12 month
Number of participants with cardiovascular death events | 1 month
Number of participants with cardiovascular death events | 3 month
Number of participants with cardiovascular death events | 6 month
Number of participants with cardiovascular death events | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Cong-xin Huang, doctor, Study Chair — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China